CLINICAL TRIAL: NCT06920992
Title: Network Mechanisms of Cognitive Control
Brief Title: Cognitive Control Functions of the Human Thalamus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Hwang (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Kai Hwang, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201808855; R01MH122613 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: Cognitive Control; Stroke; Thalamus
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Compare patients with stroke with healthy comparisons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determine the effects of subcortical thalamic lesions (Experimental): There are 3 types of testing procedures, (cognitive behavioral testing, EEG, and MRI). The types of procedures involved vary from participant to participant, depending on what kind of data investigators need and which procedure subjects agree to participate. The subject may participate in all testing procedures.
  Interventions: Behavioral: Working memory and set-switching tasks

INTERVENTIONS:
Behavioral: Working memory and set-switching tasks — A behavioral task that requires subjects to switch between stimulus- response contingencies based on a colored contextual cue. In addition, a behavioral task that requires subjects to memorize a set of visual stimuli. Subjects will then be presented with a test set and will be asked to indicate whether any stimulus therein is not part of original memorized set.

SUMMARY:
The goal of this research project is to investigate how brain lesions affect our ability to generate goal-directed behaviors - a cognitive function commonly referred to as cognitive control. To support goal-directed behaviors, the human brain must adaptively direct thoughts and actions depending on the current goals and contexts. Our principal hypothesis is that this cognitive capacity depends on a brain network architecture that can flexibly transmit, select, and inhibit information along neural pathways. Therefore, lesions and damages to critical brain network components will negatively affect behavior. To faithfully assess the structure and function of human brain networks and its disruption from brain lesions, investigators will recruit healthy adult human subjects and patients with brain lesions to participate in a multi-session study that includes cognitive behavioral tests, structural magnetic resonance imaging (MRI) using a 3 Tesla (3T) scanner, and electroencephalography (EEG) studies. During all testing sessions, subjects will perform cognitive tasks that assess their ability to select, maintain, and inhibit sensory information and generate motor responses. Their eye movements may be passively recorded during testings. 3T MRI allows for fast and high-resolution imaging of brain structures, enabling us to identify lesion loci. Investigators will use EEG to measure the electrophysiology of brain activities. All behavioral, EEG, and MRI data collected will be sent to the National Institute of Mental Health Data Archive (NDA) at the National Institute of Mental Health (NIMH).

DETAILED DESCRIPTION:
There are 3 types of testing procedures, (cognitive behavioral testing, EEG, and MRI,) that investigators will describe in detail below. The types of procedures involved vary from participant to participant, depending on what kind of data investigators need and which procedure subjects agree to participate. The subject may participate in all testing procedures, (MRI, EEG, and behavioral,) two or three. The subject is also free to decline any of the testing procedures, equivalent to not participating in the research study. For each procedure, the testing time will never exceed 3 hours, so the maximum time commitment for the subject will be 9 hrs. For each subject, no more than two testing procedures will occur within 24 hours. When two testing procedures occur within the same 24-hour period, the time between the two testing procedures will be whatever is most convenient for the subject. The time between testing procedures that do not occur within the same 24-hour period will be whatever is most convenient for the subject, (this could mean weeks or months depending on the subject.) The specific procedure(s) the subject agrees to participate in will be checked on the consent form. The order which a subject will participate in these three types of procedures will also vary from subject to subject, which depends on the subject's schedule and the availability of the research facilities.

COGNITIVE BEHAVIORAL PROCEDURES: The type of cognitive task that will be administered aimed at measuring subject's ability to monitor internal goals and intentions, maintain and manipulate information in working memory, select task-relevant information, inhibit distractions, and organize action plans to accomplish these goals. These tasks involve the presentation of visual or auditory stimuli through a computer system, and the subjects must pay attention to the presented stimuli and make button press responses. Their eye movements may be monitored by a non-invasive eye-tracking device placed 1 to 2 feet in front of the participants. The eye-tracking device passively records the subject's eye gaze direction and no part of the device will be touching the subject, therefore, there will be no negative impact on the subject's comfort. The testing time for this procedure will be 1 to 3hrs.

EEG PROCEDURES: In this procedure, subjects will have EEG recorded while concurrently monitoring behavior. Subjects are asked to sit in a testing room and have conventional EEG electrodes placed on their scalp with conducting paste. The experiments involve the presentation of images on a computer monitor, sounds through speakers or headphones. The tasks may be changed flexibly as required by our behavioral testing of the tasks (i.e., is this task too easy for subjects? Too hard? These are questions investigators can only answer once investigators begin piloting the task behaviorally), however the task will always be asking subjects to manipulate the simple or complex stimuli in mind and respond to the participants in a brief period of time. The task will get at our questions about cognitive control by engaging brain regions involved in memorizing stimuli, attending to stimuli, ignoring stimuli, and preparing responses. These are components of cognitive control that are of interest for this project. The subject is asked to respond to certain stimuli by pressing a button. All stimuli are presented at a comfortable level. Similar to the cognitive behavioral procedure, a non-invasive eye tracking device may record subject's eye movements during EEG recording. This eye-tracking device is non-invasive and no parts of the device will cause any discomfort or interfere with the EEG recording. An EEG recording session typically takes 1 to 3hrs. The subject is given breaks every 5- 10 minutes, but may request a break or stop the experiment at any time. After the testing, investigators will remove the electrodes, and provide shampoo and towels for subjects to wash off the EEG conducting paste. Investigators will provide a hairdryer.

MRI (3T) PROCEDURES: Before participants enter the magnet room, participants will be screened for contradictions (i.e., metal implant). If the subject also wears glasses that contain metal to correct their visual acuity to 20/40 or better, investigators will have the subject use plastic, MR-compatible glasses provided by the MRI center. If the subject knows their prescription it will expedite the process of finding lenses suitable for the participants. If not, a few minutes will be allocated to trying on the best fitting pair to approximate the vision required to view the screen within the MRI, which is positioned close to subjects' face. Brain anatomical MRI scans are collected. Brain anatomical MRI scans are collected to determine the location of brain structures. In MRI studies, subjects who have history of brain MRIs will be acclimated to the MRI environment in a mock scanner. This is performed at a dedicated setup at MRRF in PBDB. For comfort, foam pads are placed around the subject's head to limit head movement during the scan. A MRI scanning session takes about 40 - 60 minutes and the subject is given breaks every 5-10 minutes. The subject may request a break or stop the experiment at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults age 18-35 without neurological or psychological disorders. No metal implants. No Claustrophobia.
2. Patients with focal lesions within the thalamus. Age 18 or older. No diagnosis of psychiatric disorders. No metal implants. No Claustrophobia.
3. Patients with focal lesions that spare the frontal and parietal cortices. Age 18 or older. No diagnosis of psychiatric disorders.

No metal implants. No Claustrophobia.

Exclusion Criteria:

* claustrophobic Psychiatric conditions such as depression and ADHD. Implanted device such as cardia pacemakers and autodefbrillaotors, aneurysm, cochlear implants.
* Not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive flexibility performance as measured by accuracy, in the unit of percent of accurate responses. | 2 weeks
  Accuracy measure of the behavioral task will determine whether the hypothesized cognitive function of cognitive flexibility is impaired. Impairment will lead to below chance response.
Cognitive flexibility function as measured by reaction time to cognitive switching manipulation, un the unit of seconds. | 2 weeks
  The speed of cognitive switching can be measured by the reaction time to stimulus, in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
This is a BESH study (https://grants.nih.gov/policy-and-compliance/policy-topics/clinical-trials/besh) and the investigators will not be publishing in ICMJE journals.

REFERENCES:
- [Background] Shine JM, Lewis LD, Garrett DD, Hwang K. The impact of the human thalamus on brain-wide information processing. Nat Rev Neurosci. 2023 Jul;24(7):416-430. doi: 10.1038/s41583-023-00701-0. Epub 2023 May 26. PMID 37237103
- [Result] Cellier D, Petersen IT, Hwang K. Dynamics of Hierarchical Task Representations. J Neurosci. 2022 Sep 21;42(38):7276-7284. doi: 10.1523/JNEUROSCI.0233-22.2022. PMID 35985836
- [Result] Hwang K, Bruss J, Tranel D, Boes AD. Network Localization of Executive Function Deficits in Patients with Focal Thalamic Lesions. J Cogn Neurosci. 2020 Dec;32(12):2303-2319. doi: 10.1162/jocn_a_01628. Epub 2020 Sep 9. PMID 32902335
- [Result] Hwang K, Shine JM, Bruss J, Tranel D, Boes A. Neuropsychological evidence of multi-domain network hubs in the human thalamus. Elife. 2021 Oct 8;10:e69480. doi: 10.7554/eLife.69480. PMID 34622776
- [Result] Chen X, Leach SC, Hollis J, Cellier D, Hwang K. The thalamus encodes and updates context representations during hierarchical cognitive control. PLoS Biol. 2024 Dec 2;22(12):e3002937. doi: 10.1371/journal.pbio.3002937. eCollection 2024 Dec. PMID 39621781